CLINICAL TRIAL: NCT01489436
Title: Comparative Effectiveness of Novel Minimally Invasive Procedures
Brief Title: A Comparison of Single Port and Four Port Laparoscopic Gallbladder Removal
Acronym: CENoMIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Juliane Bingener-Casey, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-001162
Record Dates: First submitted 2011-08-25; First posted 2011-12-09 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: CHOLELITHIASIS
Keywords: gallstone disease; cholecystectomy; minimally invasive; surgical; laparoscopic; single port; cytokine
MeSH Terms: conditions — Cholelithiasis | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single port cholecystectomy (Active Comparator): In brief, a flexible, multi-sleeve 15-mm trocar designed specifically for single-port cholecystectomy will be inserted at the umbilicus via a 15-mm single incision. An additional 2-mm grasping device may be introduced in the right upper quadrant for retraction if necessary; this device is placed percutaneously without the need for a trocar. A 5-mm laparoscopic clip applier will be introduced through the periumbilical trocar to ligate the cystic artery and the cystic duct. The gallbladder will be removed through the umbilical port, adequate hemostasis is ensured, the umbilical trocar removed, and the single operative site will be closed and sterile dressings applied (four Band-Aids).
  Interventions: Procedure: Single-port cholecystectomy
- Four-port laparoscopic cholecystectomy (Active Comparator): The control procedure for the research practicum is a four-trocar laparoscopic cholecystectomy, the current gold-standard operation. This approach utilizes a 10-mm trocar placed at the umbilicus via a 15-mm incision and three separate subcostal 5-mm trocars placed via separate 5-mm incisions. The gallbladder will be removed through the umbilical trocar site. On occasion, this incision needs to be enlarged to accommodate removal of the gallbladder. Trocar sites will be closed and sterile dressings applied (four Band-Aids).
  Interventions: Procedure: Four-port laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Single-port cholecystectomy — In brief, a flexible, multi-sleeve 15-mm trocar designed specifically for single-port cholecystectomy will be inserted at the umbilicus via a 15-mm single incision. This trocar permits simultaneous introduction of multiple instruments, including a 5-mm flexible-tip laparoscope. Standard 5-mm instruments will be used for retraction and dissection. An additional 2-mm grasping device may be introduced in the right upper quadrant for retraction if necessary. A 5-mm laparoscopic clip applier will be introduced through the periumbilical trocar to ligate the cystic artery and the cystic duct. The gallbladder will be removed through the umbilical port.
  Other Names: Minimally invasive surgery
  Arms: Single port cholecystectomy
Procedure: Four-port laparoscopic cholecystectomy — The control procedure for the research practicum is a four-trocar laparoscopic cholecystectomy, the current gold-standard operation. This approach utilizes a 10-mm trocar placed at the umbilicus via a 15-mm incision and three separate subcostal 5-mm trocars placed via separate 5-mm incisions. The gallbladder will be removed through the umbilical trocar site. On occasion, this incision needs to be enlarged to accommodate removal of the gallbladder.
  Other Names: Minimally invasive surgery
  Arms: Four-port laparoscopic cholecystectomy

SUMMARY:
New minimally invasive surgical treatments are often outpatient procedures with low complication rates, promising fast recovery. The traditional physician-reported outcomes such as complication rates, blood loss, and hospital stay are not useful to guide treatment recommendations for one or the other minimally invasive procedure. This study aims to apply patient-reported outcomes developed within the NIH framework for cancer research and chronic disease treatment to the comparative effectiveness research in minimally invasive procedures for benign disease.

DETAILED DESCRIPTION:
To establish a pathway for comparative effectiveness using patient reported outcomes in minimally invasive surgery, we propose to use a readily available and easily reproducible model: cholecystectomy. Each year in the United States, approximately 750,000 patients undergo a cholecystectomy. Patients clearly prefer the laparoscopic approach over the open procedure to abdominal surgery. Initial survey data suggest that patients may also prefer even less invasive approaches.

Currently, the standard operative procedure for a patient with symptomatic gallstone disease is a laparoscopic cholecystectomy performed under general anesthesia with four small abdominal incisions. Although postoperative pain and cardiopulmonary and wound complications are much less compared to open cholecystectomy, considerable cost is generated from lost productivity in days off of work after the surgical procedure related in part to pain and the physiologic response to the stress of the operative procedure. Anecdotal data suggest that fewer incisions, especially fewer transabdominal incisions, translate into less pain, less need for narcotic pain medication and faster recovery, but randomized trial data are needed. We propose to compare the effectiveness of the novel single-port cholecystectomy with laparoscopic cholecystectomy, the current standard of care.

ELIGIBILITY:
Inclusion criteria for this study are:

1) patients undergoing cholecystectomy in an elective setting for symptomatic gallstone disease.

Exclusion criteria for the study are:

1. Patients <18 years of age
2. Pregnant patients
3. Patients with ASA-class >3
4. Patients undergoing treatment for chronic pain with opiates
5. Patients with biopsy proven gallbladder cancer
6. Patients who cannot provide consent for the study
7. Patients not willing to participate in the study
8. Prisoners/Institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | Baseline to Post Operative day 1
  The investigators will utilize the Patient-Reported Outcomes from the VAS to measure changes from Baseline to day 1 post OP. A 15-mm difference on a 100-mm visual analog scale with a standard deviation of 25 mm at any time point will constitute a clinically relevant difference.

SECONDARY OUTCOMES:
Quality of Life (QOL) | up to 7 days
  Patients QOL will be measured via Patient-Reported Outcomes Measures Information System (PROMIS) and Linear Analog Self Assessment (LASA) tools.
  PROMIS Global Health Short Form and LASA are validated assessment tools. A 2-point difference is considered the minimally important difference in chronic disease for an item in the PROMIS and LASA tools.
Heart Rate Variability (HRV) Data | During surgery from incision to closure
  HRV is the bodies' physiological response to pain as measured through digitally captured ECG combined with electronically captured blood pressure.We will measure HRV to determine subtle differences between to the two surgical approaches.
Cytokine levels in blood | Baseline, during surgery form incision to closure, 1 hour post OP and 4 hour post OP
  Frequently used biomarkers are inflammatory cytokines, specifically the serum levels of the early response pro-inflammatory cytokines TNF-α, Interleukin 1b, Interleukin 6 and Interleukin 8. We will measure and analyze these cytokine levels at set time points to determine if any subtle difference in the levels between the two surgical approaches is significant.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Bingener-Casey, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Bingener J, Skaran P, McConico A, Novotny P, Wettstein P, Sletten DM, Park M, Low P, Sloan J. A Double-Blinded Randomized Trial to Compare the Effectiveness of Minimally Invasive Procedures Using Patient-Reported Outcomes. J Am Coll Surg. 2015 Jul;221(1):111-21. doi: 10.1016/j.jamcollsurg.2015.02.022. Epub 2015 Mar 3. PMID 26095558
- See also: A Double-Blinded Randomized Trial to Compare the Effectiveness of Minimally Invasive Procedures Using Patient-Reported Outcomes. — https://www.ncbi.nlm.nih.gov/pubmed/26095558